CLINICAL TRIAL: NCT01714518
Title: Cryobiopsy vs. VATS: Efficiency and Safety in the Diagnosis of Interstitial Lung Diseases
Brief Title: Cryobiopsy vs. VATS in Diagnosis of Interstitial Lung Diseases
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Other Study IDs: WI_KryoVATS_80/2012
Record Dates: First submitted 2012-10-09; First posted 2012-10-26 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial Lung Disease; Diagnosis; Cryobiopsy; Video-assisted thoracic surgery; Lung biopsy
MeSH Terms: conditions — Lung Diseases, Interstitial; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ILD diagnosis: Patients subjected to Cryobiopsy and/or VATS for diagnosis of interstitial lung disease

SUMMARY:
The purpose of this study is to assess efficiency and safety of cryobiopsy compared to video-assisted thoracoscopic lung biopsy (VATS) in diagnosis of interstitial lung diseases (ILD). To that end, this non-interventional study prospectively collects data from patients undergoing routine diagnosis of ILD. In some of those patients less invasive diagnostic approaches do not yield a definitive diagnosis. Thus, they will ultimately be subjected to VATS if this procedure is reasonable. The information gained by this study will help to assess the significance of cryobiopsy in contrast to VATS in this particular disease group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Known or newly diagnosed interstitial lung disease (ILD)
* Indication for lung biopsy for definitive ILD diagnosis
* Informed Consent provided

Exclusion Criteria:

* Age < 18 years
* Inability or contraindication to undergo any form of invasive diagnostic procedure associated with diagnosis of interstitial lung disease
* Severely restricted CO diffusion capacity (<50%)
* Pregnancy, lactation
* Any medical, psychological or other condition restricting the patient's ability to provide informed consent
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients undergoing routine diagnosis of known or suspected interstitial lung disease
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-10-16 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of diagnostic cryobiopsies | up to 3 days
  For the individual study participant, the result of the cryobiopsy (whether it is diagnostically helpful, i.e. "diagnostic" or not, i.e. "inconclusive") will be documented when it is available, which will be within 3 days. The overall number of diagnostic cryobiopsies will be calculated once the study is complete.

SECONDARY OUTCOMES:
Rate of complications during cryobiopsy | During and up to 48 hours after procedure
  Number of complications associated with cryobiopsy, divided into three categories of severity: mild/moderate/severe
Rate of complications during VATS | During and up to 10 days after procedure
  Number of complications associated with VATS, divided into three categories of severity: mild/moderate/severe

CONTACTS AND LOCATIONS:
Locations (1):
- Bethanien Hospital, Clinic for Pneumology and Allergology, Center for Sleep and Respiratory Medicine, Solingen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Ryu JH, Olson EJ, Midthun DE, Swensen SJ. Diagnostic approach to the patient with diffuse lung disease. Mayo Clin Proc. 2002 Nov;77(11):1221-7; quiz 1227. doi: 10.4065/77.11.1221. PMID 12440558
- [Background] Collard HR, King TE Jr. Demystifying idiopathic interstitial pneumonia. Arch Intern Med. 2003 Jan 13;163(1):17-29. doi: 10.1001/archinte.163.1.17. PMID 12523913
- [Background] King TE Jr. Clinical advances in the diagnosis and therapy of the interstitial lung diseases. Am J Respir Crit Care Med. 2005 Aug 1;172(3):268-79. doi: 10.1164/rccm.200503-483OE. Epub 2005 May 5. PMID 15879420
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Ferson PF, Landreneau RJ, Dowling RD, Hazelrigg SR, Ritter P, Nunchuck S, Perrino MK, Bowers CM, Mack MJ, Magee MJ. Comparison of open versus thoracoscopic lung biopsy for diffuse infiltrative pulmonary disease. J Thorac Cardiovasc Surg. 1993 Aug;106(2):194-9. PMID 8341061
- [Background] Miller JD, Urschel JD, Cox G, Olak J, Young JE, Kay JM, McDonald E. A randomized, controlled trial comparing thoracoscopy and limited thoracotomy for lung biopsy in interstitial lung disease. Ann Thorac Surg. 2000 Nov;70(5):1647-50. doi: 10.1016/s0003-4975(00)01913-5. PMID 11093503
- [Background] Ayed AK, Raghunathan R. Thoracoscopy versus open lung biopsy in the diagnosis of interstitial lung disease: a randomised controlled trial. J R Coll Surg Edinb. 2000 Jun;45(3):159-63. PMID 10881481
- [Background] Bensard DD, McIntyre RC Jr, Waring BJ, Simon JS. Comparison of video thoracoscopic lung biopsy to open lung biopsy in the diagnosis of interstitial lung disease. Chest. 1993 Mar;103(3):765-70. doi: 10.1378/chest.103.3.765. PMID 8449066
- [Background] Babiak A, Hetzel J, Krishna G, Fritz P, Moeller P, Balli T, Hetzel M. Transbronchial cryobiopsy: a new tool for lung biopsies. Respiration. 2009;78(2):203-8. doi: 10.1159/000203987. Epub 2009 Feb 21. PMID 19246874
- [Background] Pajares V, Torrego A, Puzo C, Lerma E, Gil De Bernabe MA, Franquet T. [Transbronchial lung biopsy using cryoprobes]. Arch Bronconeumol. 2010 Mar;46(3):111-5. doi: 10.1016/j.arbres.2009.09.012. Epub 2009 Nov 25. Spanish. PMID 19939546
- [Background] Aktas Z, Gunay E, Hoca NT, Yilmaz A, Demirag F, Gunay S, Sipit T, Kurt EB. Endobronchial cryobiopsy or forceps biopsy for lung cancer diagnosis. Ann Thorac Med. 2010 Oct;5(4):242-6. doi: 10.4103/1817-1737.69117. PMID 20981186
- [Background] Hetzel J, Eberhardt R, Herth FJ, Petermann C, Reichle G, Freitag L, Dobbertin I, Franke KJ, Stanzel F, Beyer T, Moller P, Fritz P, Ott G, Schnabel PA, Kastendieck H, Lang W, Morresi-Hauf AT, Szyrach MN, Muche R, Shah PL, Babiak A, Hetzel M. Cryobiopsy increases the diagnostic yield of endobronchial biopsy: a multicentre trial. Eur Respir J. 2012 Mar;39(3):685-90. doi: 10.1183/09031936.00033011. Epub 2011 Aug 18. PMID 21852332
- [Derived] Hagmeyer L, Theegarten D, Wohlschlager J, Hager T, Treml M, Herkenrath SD, Hekmat K, Heldwein M, Randerath WJ. Transbronchial cryobiopsy in fibrosing interstitial lung disease: modifications of the procedure lead to risk reduction. Thorax. 2019 Jul;74(7):711-714. doi: 10.1136/thoraxjnl-2018-212095. Epub 2019 Mar 9. PMID 30852561
- [Derived] Hagmeyer L, Theegarten D, Treml M, Priegnitz C, Randerath W. Validation of transbronchial cryobiopsy in interstitial lung disease - interim analysis of a prospective trial and critical review of the literature. Sarcoidosis Vasc Diffuse Lung Dis. 2016 Mar 29;33(1):2-9. PMID 27055830